CLINICAL TRIAL: NCT07315659
Title: Time-Restricted Eating as a Potential Strategy to Promote Weight Loss Maintenance in Patients With Obesity (REGANE)
Brief Title: Time-Restricted Eating as a Potential Strategy to Promote Weight Loss Maintenance in Patients With Obesity
Acronym: REGANE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Clinico Universitario San Cecilio (Other); University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Guillermo Sanchez Delgado, Ramon y Cajal Researcher (Tenure-track position), Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSD-2024-003
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Obesity; Calorie restriction; Intermittent Fasting; Weight loss; Weight loss maintenance; Weight regain; Time-restricted eating; Diet
MeSH Terms: conditions — Obesity; Intermittent Fasting; Weight Loss | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (eating within 8 hours/day or less) (Experimental): Participants in the time-restricted eating group will be instructed to concentrate all daily meals to 8 hours or less
  Interventions: Behavioral: Calorie restriction (Dietary intervention); Behavioral: Time-restricted eating
- Regular eating window (eating within 12 hours/day or more) (Sham Comparator): Participants in the regular eating group will be instructed to spread all daily meals within a of 12 hours or more.
  Interventions: Behavioral: Calorie restriction (Dietary intervention); Behavioral: Regular eating window

INTERVENTIONS:
Behavioral: Calorie restriction (Dietary intervention) — Calorie restriction intervention consisting on a meal plan designed to induce an 8-10% weight loss over a 12-16 week period.
Behavioral: Regular eating window — Receiving instructions to maintain their regular eating window (12h/d or more) both during the 12-16 weeks of calorie restriction and the 12 months following its completion.
  Arms: Regular eating window (eating within 12 hours/day or more)
Behavioral: Time-restricted eating — Receiving instructions to confine all daily meals to a period of 8 hours or less (at least 6 days a week) both during the 12-16 weeks of calorie restriction and the 12 months following its completion.
  Arms: Time-restricted eating (eating within 8 hours/day or less)

SUMMARY:
While body weight reduction can be achieved through various interventions in people living with obesity, most patients regain a substantial proportion of the lost weight within the following months. There is a lack of effective interventions to prevent this regain, making weight regain one of the most pressing challenges in obesity management. The goal of this clinical trial is to determine whether adhering to time-restricted eating (TRE; a form of intermittent fasting) during and after a dietary weight loss intervention, promotes weight maintenance to a greater extent than consuming all daily meals within 12 hours or more. Additionally, the study will address other questions, such as whether TRE improves body composition, insulin sensitivity, and cardiometabolic risk factors; whether the TRE intervention produces effects on different components of energy balance or related behaviors; and whether prior exposure to the TRE intervention influences eating window duration and weight change over the subsequent 24 months.

The study will compare participants who concentrate all their food intake within 8 hours or less with those who consume all their daily meals within 12 hours or more. All participants will follow a calorie-restricted diet designed to induce an 8-10% weight loss over 12-16 weeks and will be followed for several months after the weight loss intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index of 30-45 kg/m2.
* Have safety laboratory test results (general biochemistry and complete blood count) within the normal reference range or with abnormalities considered clinically insignificant by the medical research team and that do not require the initiation of drug treatment.
* Have sufficient venous access for the blood sampling required by the procedures described in this protocol, and not have a phobia of needles or blood.
* Maintain a usual intake window of 12 hours or longer at least 5 days a week and have a response rate greater than 85% during the self-recording carried out during the screening process.
* Willingness and ability to consume all foods provided during the outcome assessment and dietary intervention.
* Being able to understand and undergo the procedures that are part of the study, in the opinion of the research team.
* Availability to participate in the study.
* Be willing to complete the study regardless of the group to which they are assigned.

Exclusion Criteria:

* Having received a diagnosis or presenting signs or symptoms that, in the opinion of the research team, could contraindicate TRE intervention or any of the procedures included in the study.
* Having been diagnosed with or having a history of metabolic (including a diagnosis of any type of diabetes mellitus), hematological, pulmonary, cardiovascular, gastrointestinal, neurological, immune, hepatic, renal, urological or psychiatric diseases that could interfere with the study results or compliance with the protocol.
* Having undergone any surgical procedure that, in the opinion of the research team, could alter energy metabolism or digestive function during the course of the study.
* Taking drugs or supplements that are likely to alter body weight or appetite.
* Have experienced weight loss of more than 10% in the last two years, or more than 5% in the last 6 months, unless all the weight lost has been regained.
* Follow unconventional eating patterns, such as vegan or fasting diets, or be unable to tolerate the foods provided during the study.
* Being pregnant or planning to become pregnant within the next two years.
* Being in the postpartum phase (within 12 months of giving birth) or breastfeeding.
* Being in the perimenopausal stage, defined as meeting the criteria of irregular menstrual cycles, hormonal changes indicative of perimenopause, or the presence of menopausal symptoms.
* Participating in a nutritional intervention or treatment or having done so during the previous 3 months.
* Having been diagnosed with or showing signs or risk factors for the development of an eating disorder.
* Experiencing frequent interruptions in the sleep-wake cycle.
* Having clinically significant gastric emptying abnormalities, a current diagnosis of any form of diabetes, blood pressure greater than 160/90 mm Hg, or heart rate below 50 or above 100 beats per minute (sitting), with or without stable doses of antihypertensive medication.
* Have an active or untreated malignant disease or be in remission from a clinically significant malignant disease for less than five years prior to the time of evaluation.
* Having a history of drug or alcohol abuse or testing positive for drugs, unless due to medication prescribed by a healthcare professional.
* Smoking, vaping, or regular use of tobacco products, unless there have been periods of at least 24 consecutive hours without consumption during the last 4 weeks.
* Regular consumption of caffeine in excess of the equivalent of 3 espressos per day (225 mg/day).
* Being a direct relative or cohabitant of research team personnel.
* Any other condition that, in the opinion of the research team, makes participation in the study inadvisable.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in weight (Kg) during the 6 months following the end of the calorie restriction intervention | 6 after the end of the dietary intervention - End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss).

SECONDARY OUTCOMES:
Weight (Kg) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention
Waist circumference (cm) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Hip Circumference (cm) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fat mass (kg) by DXA | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fat free mass (kg) by DXA | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fat mass (kg) by Bioimpendaciometry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fat free mass (kg) by Bioimpendaciometry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Body Mass Index (kg/m2) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Resting Energy Expenditure (kcal/day) measured by indirect calorimetry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Posprandial Energy Expenditure (kcal/day) measured by indirect calorimetry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Fasting nutrient utilization rates (g/min) measured by indirect calorimetry and protein excretion | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Postprandial nutrient utilization rates (g/min) measured by indirect calorimetry and protein excretion | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Energy Intake (kcal) in an Ad-Libitum Meal Test | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Energy efficiency (W/KJ) while cycling, assessed by indirect calorimetry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Maximal fat oxidation (g/min) by indirect calorimetry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Physical activity (counts/day) measured by accelerometry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 after the end of dietary intervention.
Sedentary time (min/day) measured by accelerometry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention
Habitual food consumption collected by a food frecuency questionnaire | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Serum Total Cholesterol (mg/dl) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum LDL cholesterol (mg/dl) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum HDL cholesterol (mg/dl) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum triglycerides (mg/dl) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum glucose (mg/dl) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum insulin (U/ml) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum hemoglobin A1c (mmol/mol) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum thyrotropin (µU/mL) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum Alanine Transaminase (U/L) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention
Serum Aspartate Transaminase (U/L) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum gamma-glutamyl transferase (U/L) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Serum C-reactive protein (mg/dL) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Craving Control measured using the Control of Eating Weekly Questionnaire (CoEQ) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Positive Mood measured using the Control of Eating Weekly Questionnaire (CoEQ) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Craving for Sweet Foods measured using the Control of Eating Weekly Questionnaire (CoEQ) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Craving for Savory Foods measured using the Control of Eating Weekly Questionnaire (CoEQ) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fasting appetite-related sensations measured using "Visual Analogue Scales (VAS)" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Meal-induced changes in appetite-related sensations measured using "Visual Analogue Scales (VAS)" in response to a meal | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Fasting Liking and Wanting measured using Leeds Food Preference Questionnaire | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Liking and Wanting in response to a meal measured using Leeds Food Preference Questionnaire | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Meal-induced changes in serum glucose concentration (mg/dL) in response to a standardized meal | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Meal-induced changes in serum insulin concentration (U/ml) in response to a standardized meal | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Cognitive restriction of food intake measured using the "Three-Factor Eating Questionnaire" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Food disinhibition measured using the "Three-Factor Eating Questionnaire" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Subjective hunger measured using the "Three-Factor Eating Questionnaire" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Binge eating behavior measured using the "Binge Eating Questionnaire" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Sleep time (min) measured by accelerometry | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Handgrip strength (kg) measured using a dynamometer | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Functional mobility measured by "Timed Up and Go (TUG)" test | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Walking speed (m/s) measured by a gait speed test | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Independence in activities of daily living (ADL) measured by "Barthel Index" | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention
Food cravings measured using the "Food Craving Inventory" questionnaire | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention
Carbohydrate intake (g/day) collected through three 24-hour recalls | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fat intake (g/day) collected through three 24-hour recalls | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Protein intake (g/day) collected through three 24-hour recalls | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Fiber intake (g/day) collected through three 24-hour recalls | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Changes in appetite-related sensations measured using "Visual Analogue Scales (VAS)" in response to a submaximal stress test | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 6 months after the end of dietary intervention.
Resting heart rate variability | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Resting Systolic blood pressure (mmHg) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.
Resting Diastolic blood pressure (mmHg) | Baseline; End of dietary intervention (Week 12/16, depending on achievement of 8-10% weight loss); 1, 3, 6, 12, 18, 24 and 36 months after the end of dietary intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiology, Faculty of Medicine, University of Granada., Granada, Granada, Spain